CLINICAL TRIAL: NCT05296694
Title: Predictors of In-hospital MORtality in CORonary Care Patients in TURKey
Brief Title: Mortality Predictors in Coronary Care in Turkey
Acronym: MORCOR-TURK
Status: Completed | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, İbrahim Ersoy, MD, Assistant Professor, Afyonkarahisar Health Sciences University
Other Study IDs: 3450
Record Dates: First submitted 2022-03-08; First posted 2022-03-25 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Death, Cardiac
Keywords: Coronary Care Unit; Mortality; Predictors
MeSH Terms: conditions — Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Care Patients: All patients admitted to coronary care unit with cardiovascular diseases.

SUMMARY:
This study was undertaken to investigate and document the mortality rates and predictors in coronary care unit (CCU) patients in Turkey.

It is designed to be a multicenter, observational, cross-sectional, and descriptive study. It will be conducted in 50 centers in 12 regions of Turkey. The study does not include any interventional or treatment procedures.

At the end of the study, clinicians will have up-to-date information about predictors of mortality in CCU patients.

DETAILED DESCRIPTION:
The MORCOR-TURK study will be conducted as a nationwide registry in 50 tertiary cardiology centers selected from each EuroStat NUTS region in Turkey according to their population sample weight, prioritizing the volume of hospitals in each region. All consecutive patients admitted to the coronary care units (CCU) will be prospectively admitted during a predefined period of 1 month. The study will be conducted by cardiologists in hospitals who regularly treat cardiac patients. Led by the Cardiology Department of Kutahya Evliya Celebi Research and Training Hospital, 50 centers will be included in the study.

There has not been any large-scale epidemiological study on coronary care patients in Turkey recently. Therefore, up-to-date information in this group of patients is lacking. In particular, significant reductions in mortality and morbidity are expected, thanks to improved medical and interventional facilities. In the light of current data, the investigators designed a large-scale study to document mortality rates and predictors in CCU patients.

In this study, the investigators will include consecutive patients admitted to CCU with cardiovascular indications in all participating centers. Patients will be followed and treated by experienced cardiologists and no further experimental intervention will be planned. In the first part of the study, the investigators will record in-hospital mortality rates and try to identify the best predictors. In the second part of the MORCOR-TURK trial which will have a cohort design, the investigators will follow the successfully discharged patients for 1 year. At the end of the follow-up, investigators will assess the risk factors and predictors of cardiovascular events as secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* hospitalized with cardiovascular diseases
* individuals (or relatives for unconscious patients) who gave written informed consent

Exclusion Criteria:

* younger than 18 years of age
* rejecting to sign an informed consent
* hospitalized to CCU by other departments with noncardiac indications
* patients with active severe noncardiac chronic disease (chronic obstructive pulmonary disease, systemic diseases, and malignancy)
* no vital signs despite adequate cardiopulmonary resuscitation during hospitalization
* rejected to stay in CCU and discharged with his/her own request

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients (age≥18) admitted to the coronary intensive care unit for cardiovascular reasons in all centers participating in the study between the dates specified.
Sampling Method: Non-Probability Sample
Enrollment: 2560 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
All cause mortality | In-hospital (up to two-weeks)
  All types of mortality in-hospital follow up

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Kahraman, MD, Study Director — Kutahya Health Sciences University Evliya Celebi Research and Training Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Afyonkarahisar Health Sciences University, Afyonkarahisar
  - Kutahya Evliya Celebi Research and Training Hospital, Kütahya

REFERENCES:
- [Background] Ratcliffe JA, Wilson E, Islam S, Platsman Z, Leou K, Williams G, Lucido D, Moustakakis E, Rachko M, Bergmann SR. Mortality in the coronary care unit. Coron Artery Dis. 2014 Jan;25(1):60-5. doi: 10.1097/MCA.0000000000000043. PMID 24121428
- [Background] Filizcan U, Kurc E, Cetemen S, Soylu O, Aydogan H, Bayserke O, Yilmaz M, Uyarel H, Ergelen M, Orhan G, Ugurlucan M, Eren E, Yekeler I. Mortality predictors in ST-elevated myocardial infarction patients undergoing coronary artery bypass grafting. Angiology. 2011 Jan;62(1):68-73. doi: 10.1177/0003319710369103. Epub 2010 May 12. PMID 20462895
- [Background] Hayiroglu MI, Keskin M, Uzun AO, Yildirim DI, Kaya A, Cinier G, Bozbeyoglu E, Yildirimturk O, Kozan O, Pehlivanoglu S. Predictors of In-Hospital Mortality in Patients With ST-Segment Elevation Myocardial Infarction Complicated With Cardiogenic Shock. Heart Lung Circ. 2019 Feb;28(2):237-244. doi: 10.1016/j.hlc.2017.10.023. Epub 2017 Nov 14. PMID 29191504
- [Background] Campanile A, Castellani C, Santucci A, Annunziata R, Tutarini C, Reccia MR, Del Pinto M, Verdecchia P, Cavallini C. Predictors of in-hospital and long-term mortality in unselected patients admitted to a modern coronary care unit. J Cardiovasc Med (Hagerstown). 2019 May;20(5):327-334. doi: 10.2459/JCM.0000000000000785. PMID 30865139
- [Derived] Taylan G, Kaya C, Ozbek M, Kurt F, Kacmaz Y, Akkaya F, Kahraman F, Yilmaz AS. Short-Term Prognosis of Elderly Patients Admitted to the Coronary Care Unit: A Subgroup Analysis of the MORCOR-TURK (Mortality and Morbidity in Coronary Care Units in Turkiye) Trial. Turk Kardiyol Dern Ars. 2024 Sep;52(6):411-419. doi: 10.5543/tkda.2024.51282. PMID 39225647
- [Derived] Kahraman F, Ersoy I, Yilmaz AS, Atici A, Tekin AM, Acar B, Kaya C, Kara F, Kurt F, Avci Demir F, Cerik IB, Yilmaz I, Adali MK, Yeni M, Tascanov MB, Yenercag M, Sahin M, Duz R, Gulasti S, Omur SE, Topuz S, Hidayet S, Kacmaz Y, Aygul N. Rationale, Design, and Methodology of the MORCOR-TURK Trial: Predictors of In-hospital MORtality in CORonary Care Patients in Turkey. Anatol J Cardiol. 2023 May;27(5):258-265. doi: 10.14744/AnatolJCardiol.2022.2824. PMID 37119186